CLINICAL TRIAL: NCT07281690
Title: Enhancing Skin Rejuvenation A Single-Blind, Randomized Control Study on the Combined Efficacy of Aerolase 1064 nm YAG Laser and Exosomes Derived From Umbilical Cord Mesenchymal Stem Cells
Brief Title: Enhancing Skin Rejuvenation Using Laser and Exosomes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laser Beamer Skincare (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-08-089-2058
Record Dates: First submitted 2025-10-27; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-10

CONDITIONS: Laser Therapy; Exosomes

STUDY DESIGN:
Intervention Model Description: Subjects receive lasering on their entire face and apply exosomes to a randomly assigned side of one side of their face. 3 laser sessions and 60 days of exosomes applied daily.
Masking Description: Participants were aware of the side of the intervention, but the investigator performing outcome assessments and data analysis was masked, meaning the subjects applied the exosomes to the side of the face that was randomly assigned by drawing a ticket with a de-idenifying number and L or R-the side the exosomes were to be applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Split-Faced Design) (Experimental): All participants received a 1064-nm Nd:YAG laser treatment to the entire face. Exosomes (UC-MSC-derived topical serum) were applied only to the randomly assigned side of the face.
  The opposite side received laser only.
  Interventions: Device: 1064-nm Nd:YAG Laser Treatment; Biological: Topical Umbilical Cord-Derived Exosomes (UC-MSC Exosomes)

INTERVENTIONS:
Device: 1064-nm Nd:YAG Laser Treatment — A non-ablative 1064-nm Nd:YAG laser (Aerolase Neo Elite) delivered to the entire face at each treatment visit.
Biological: Topical Umbilical Cord-Derived Exosomes (UC-MSC Exosomes) — Description:
  Topical application of a laboratory-processed umbilical cord lining mesenchymal stem-cell-derived exosome serum.
  Applied twice daily to the randomly assigned half of the face for 60 days following each laser session.
  Other Name: Exosome serum; UC-MSC exosome solution.

SUMMARY:
Enhancing Skin Rejuvenation A Single-Blind, Randomized Control Study on the Combined Efficacy of Aerolase 1064 nm YAG Laser and Exosomes Derived from Umbilical Cord Mesenchymal Stem Cells

DETAILED DESCRIPTION:
1. Brief Summary This study evaluates the combined efficacy of the Aerolase 1064-nm Nd:YAG laser and umbilical cord-derived mesenchymal stem cell (UC-MSC) exosomes for skin rejuvenation. The investigation uses a single-blind, randomized, split-face design to compare laser alone versus laser plus topical exosomes. Participants undergo facial analysis, laser treatment, and structured follow-up assessments to measure changes in skin redness, wrinkles, spots, tone, and overall skin quality.
2. Detailed Description Detailed Description The study is conducted in Wichita, Kansas, a city of approximately 400,000 residents. Women constitute roughly 50% of the population, with an estimated one-third between ages 45-70. The percentage needed for this study represents less than 1% of the target demographic. Recruitment begins after IRB approval, with approximately 20 hours per week devoted to screening, enrolling, treating, and evaluating participants.

All study procedures occur at a single clinical site. The Principal Investigator (PI) is responsible for all recruitment, study activities, laser treatments, data entry, and follow-up coordination. The PI has over 30 years of nursing experience, including extensive clinical practice in women's health and mental health. Two additional nurse practitioners are available for consultation in case of medical concerns.

Participants are provided with study-related materials, including a consent form, PRO-X exosome information, a study protocol handout, and sunscreen. Eligible participants undergo baseline 3D HALO facial analysis and the initial Aerolase laser treatment. Participants draw a randomized ticket indicating "L" or "R," determining which facial side receives exosome application. The PI remains blinded to the allocation throughout the study.

Follow-up visits occur on Days 30, 45, and 60, with automated reminders sent via the clinic scheduling platform. Participants may contact the study site at any time with questions or concerns.

* Number of Subjects Twenty female participants are recruited from the Wichita metropolitan area. A minimum of ten participants is considered acceptable for study viability. All study visits occur at a single site.
* Recruitment Methods Recruitment uses flyers, social media posts, the clinic's website, Google business page, and professional networking meetings. Interested individuals contact the study site through phone, email, text message, or online scheduling. Eligibility screening includes verification of age and availability for the full study period.
* Study Duration Total participation time ranges from 60-80 days. Follow-up windows allow for minor scheduling adjustments. Total enrollment is expected to take 3-4 weeks, with full study completion-including data analysis-estimated at 180 days.
* Procedures Involved

  1. Standardized skin evaluation questionnaire on Days 1, 30, 45, and 60.
  2. HALO 3D facial imaging on Days 1, 30, 45, and 60.
  3. Aerolase 1064-nm Nd:YAG laser treatment to the full face at each visit.
  4. Randomized assignment of exosome application to either the left or right facial side.
  5. Twice-daily exosome application at home on the assigned side.
  6. Daily sunscreen use on the full face for the duration of the study. The study design is a single-blind, randomized, controlled, interventional trial evaluating changes in key skin parameters, including moisture, laxity, wrinkles, pigmentation, texture, tone, radiance, and pore size.

HALO Analyzer devices automatically calibrate before each session, ensuring consistency in measurement. Identical photographic conditions are maintained across all time points.

Laser treatments follow Aerolase manufacturer guidelines tailored to Fitzpatrick skin type. The PI is trained in all device operations, ensuring standardization across sessions.

14) Data Management Objective data are collected through the HALO Analyzer and stored under de-identified subject numbers. Paired t-tests are used to compare pre- and post-treatment values for each facial side. The paired design accounts for within-subject variability.

Data verification includes cross-checking HALO outputs with participant self-assessments. Photographic documentation is reviewed immediately after capture to ensure clarity.

14.2 Confidentiality and Data Security All participant data-including photographs and self-assessments-are stored on a password-protected computer in a locked office. De-identified numeric codes replace participant names after enrollment. Only the PI and designated blinded nurse practitioner raters have access to study data.

Data will be securely retained for three years.

* Protecting Privacy of Subjects Participants are assigned a unique study number upon enrollment. All study forms, HALO images, and assessments are stored under this number. Only the PI has access to identifying information required for scheduling or follow-up communication. Nurse practitioner raters evaluate photos labeled with de-identified numbers only.
* Future Use of Data De-identified data will be maintained for three years and may be used for scientific publication or future research analyses as stated in the consent. No identifiable information will be released.
* Ensuring Safety of Subjects Risks are minimal and may include transient redness or irritation from the laser or topical products.
* Withdrawal of Subjects Participants may withdraw at any time for scheduling or personal reasons. Withdrawal reasons will be documented when possible. Data from participants who withdraw prior to completing the study will not be included in the final analysis.

ELIGIBILITY:
Inclusion Criteria:

* Females between the ages of 45-70

Exclusion Criteria:

* Women who are pregnant

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female at birth
Enrollment: 20 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
Title: Mean Change in Nurse-Photographic Rating Scores Between Exosome-Treated and Control Sides | 60 days
  Primary Outcome Measure 1
  Description:
  This outcome measures the difference between the exosome-treated and control sides using independent evaluations by three nurse practitioners. Ratings are scored on a 1-3 scale (1 = left side better, 2 = right side better, 3 = no difference).
  Time Frame: Day 60 Scoring Interpretation: Higher values indicate greater improvement on the exosome-treated side.

SECONDARY OUTCOMES:
Title: Mean Change in HALO Image Pro 3D Analyzer Scores (Redness, Wrinkles, Pigmentation, Tone) | 60 days
  Primary Outcome Measure 2
  Description:
  This outcome measures changes in HALO imaging parameters (redness, wrinkles, pigmentation, and tone) between the exosome-treated and control sides.
  Time Frame: Day 30 and Day 60 Scoring Interpretation: Higher scores represent greater improvement.

OTHER OUTCOMES:
Title: Mean Change in FACE-Q Appearance Appraisal Scores Between Exosome-Treated and Control Sides | 60 days
  Primary Outcome Measure 3
  Description:
  The FACE-Q Appearance Appraisal module includes 11 items scored from 1-4. Minimum = 1, Maximum = 4. Higher scores indicate improvement. Per-subject mean scores are calculated and compared between sides from baseline to follow-up.
  Time Frame: Day 30, Day 45, Day 60 Scoring Interpretation: Higher change scores represent greater patient-perceived improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- LaserBeamerSkincare, Wichita, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) from this study will not be shared. The dataset includes small-sample photographic images and FACE-Q responses that cannot be fully de-identified without compromising participant privacy. In addition, the study was not designed with external data sharing as a planned component.